CLINICAL TRIAL: NCT03310749
Title: A Randomized, Open-label, Multiple Dosing, Three-way Crossover Clinical Trial to Investigate the Pharmacokinetic Drug-drug Interaction of Gemigliptin and Metformin After Oral Administration in Healthy Mexican Male Subjects
Brief Title: An Assessment of Pharmacokinetic Gemigliptin and Metformin Interactions in Healthy Mexican Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stendhal Americas, S.A. (Industry)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG/STDHL-DPCL009bis
Record Dates: First submitted 2017-09-13; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus; DPP-IV inhibitor; Drug-Drug Interactions; Ethnicity
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444; Metformin

STUDY DESIGN:
Intervention Model Description: Open, randomized, multiple dose, three way, three period, cross over, drug-drug interaction, safety and tolerability study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment sequence A (Other): Gemigliptin 50 mg q.d. during 7 days, metformin 1000 mg twice a day during 7 days and gemigliptin 50 mg q.d + metformin 1000 mg twice a day during 7 days.
  Interventions: Drug: Gemigliptin; Drug: Gemigliptin 50 mg q.d. + metformin 1000 mg twice a day; Drug: Metformin
- Treatment sequence B (Other): Gemigliptin 50 mg q.d + metformin 1000 mg twice a day during 7 days, gemigliptin 50 mg q.d. during 7 days, metformin 1000 mg twice a day during 7 days
  Interventions: Drug: Gemigliptin; Drug: Gemigliptin 50 mg q.d. + metformin 1000 mg twice a day; Drug: Metformin
- Treatment sequence C (Other): Metformin 1000 mg twice a day during 7 days, gemigliptin 50 mg q.d + metformin 1000 mg twice a day during 7 days, gemigliptin 50 mg q.d. during 7 days
  Interventions: Drug: Gemigliptin; Drug: Gemigliptin 50 mg q.d. + metformin 1000 mg twice a day; Drug: Metformin

INTERVENTIONS:
Drug: Gemigliptin — A 7-day treatment period with gemigliptin 50 mg q.d., followed by a 5-day washout period; a 7 day treatment period with metformin 1000 mg twice a day followed by a 5-day washout period and a final 7-day treatment period with gemigliptin 50 mg q.d. + metformin 1000 mg twice a day
  Other Names: Metformin; Gemigliptin 50 mg q.d. + metformin 1000 mg twice a day
Drug: Gemigliptin 50 mg q.d. + metformin 1000 mg twice a day — A 7-day treatment period with gemigliptin 50 mg q.d. + metformin 1000 mg twice a day followed by a 5-day washout period; a 7-day treatment period with gemigliptin 50 mg q.d. followed by a 5-day washout period and a final 7-day treatment period with metformin 1000 mg twice a day
  Other Names: Gemigliptin; Metformin
Drug: Metformin — A 7-day treatment period with 1000 mg metformin twice a day followed by a 5-day washout period; a 7-day treatment period with gemigliptin 50 mg q.d.+ metformin 1000 mg twice a day followed by a 5-day washout period and a final 7-day treatment period with gemigliptin 50 mg q.d.
  Other Names: Gemigliptin 50 mg q.d. + metformin 1000 mg twice a day; Gemigliptin

SUMMARY:
This is an open, randomized (randomization ratio: 1:1), multiple dose, three way, three period cross over study to assess the potential for drug drug interactions between gemigliptin (a DPP-IV inhibitor mainly metabolized by CYP3A4) and metformin in a sample of healthy Mexican volunteers, aimed to determine whether the observed lack of drug-drug interactions between gemigliptin and metformin in the Korean population is reproducible in an ethnically different population characterized by a significant difference in the frequency of CYP3A4 polymorphisms associated with decreased enzymatic activity, such as CYP3A4*1b, in comparison with Asian populations.

DETAILED DESCRIPTION:
Consenting, eligible healthy adult subjects sequentially received either gemigliptin 50 mg q.d., metformin 1000 mg twice a day or gemigliptin 50 mg q.d. plus metformin 1000 mg twice a day during 3 consecutive 7 day treatment periods separated by two 5-day washout intervals, in accordance with a randomly assigned treatment sequence. Starting on the sixth treatment period day, participating subjects underwent safety assessments and repeated (24 hour) blood and urine sampling for pharmacokinetic analysis. All subjects attended to a post-study visit for final safety assessments within 8 days of study completion or early withdrawal.

Urine and plasma samples where processed to determine gemigliptin and metformin concentrations using validated analytical methods and pharmacokinetic profiles of both gemigliptin and metformin were obtained using a non-compartmental method; both the rate and degree of gemigliptin and metformin absorption resulting from their concomitant administration relative to the administration of each drug alone were assessed in search of potential pharmacokinetic interactions, Finally, a post hoc assessment of the degree and rate of the absorption of gemigliptin in the study population relative to those of a group of Korean subjects participating in phase I, repeated dose gemigliptin studies was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects at age between 20 and 45 at the screening test
* Subjects with a body weight of 55kg or more but less than 90kg and a Body Mass Index (BMI) of between 18.0 or more but less than 27.0

  * BMI (kg/m2) = Weight (kg) / {Height (m)}2
* Subjects who show the blood glucose level within the range of 70-125 mg/dL at the fasting plasma glucose (FPG) test conducted at screening
* Subjects who fully understand this clinical trial after hearing a detailed explanation about it, make a decision to participate in it by his/her own free will, and sign an informed consent form to comply with the precautions

Exclusion Criteria:

* Subjects who have a present condition or past history of any disease involving liver, kidney, nervous system, immune system, respiratory system, or endocrine system, hematologic and oncologic disease, cardiovascular disease, or psychiatric disorder (mood disorder, obsessive-compulsive disorder, etc.) (including subjects carrying hepatitis virus in case of liver disease)
* Subjects with a past history of a gastrointestinal system disease (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or a gastrointestinal system surgery (however, subjects with a history of appendectomy or hernioplasty are not excluded)
* Subjects with a medical history of allergic reaction to drugs (aspirin, antibiotics, etc.) or clinically significant hypersensitivity reaction
* Subjects who show one of the following results at screening test:

  * Exceeds 1.5 times the upper limit of the normal range of blood AST (SGOT) and ALT (SGPT)
  * The creatinine clearance calculated by Cockcroft-Gault equation is below 80 mL/min.
  * QTc > 450 ms in ECG or clinically significant abnormal rhythm
* In the vital signs measured in sitting position after a rest for 3 minutes or longer, subjects who showed a systolic blood pressure of ≤ 100 mmHg or ≥ 150 mmHg, or a diastolic blood pressure of ≤ 60 mmHg or ≥ 95 mmHg)
* Subjects who have a past history of drug abuse or have shown a positive reaction to drugs that are used in abusive manner or cotinine at a urine drug screening
* Subjects who have taken any ethical drug or an herbal medication within 2 weeks before the date of first administration or have taken any over-the-counter (OTC) drug or vitamin preparation within 1 week (however, they can be included as subjects if considered appropriate at the investigator's discretion judgment)
* Subject who have already participated in other clinical trials within 2 months before the date of first drug administration
* Subject who have had whole blood donation within 2 months or component blood donation within 1 month before the date of first drug administration, or transfusion in 1 month before the date of first drug administration
* Subjects who have been drinking alcohol continuously (more than 21 units/week, 1 unit = 10 g of pure alcohol) or can't refrain from drinking alcohol during the clinical trial period
* Smokers (however, if the subject stopped smoking more than 3 months before the date of the first drug administration, he/she can be selected as a subject)
* 12) Subjects who have had grapefruit/ any food containing caffeine within 3 days before the date of the first drug administration

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2016-05-03 (Actual)

PRIMARY OUTCOMES:
Gemigliptin AUCτ,ss Geometric Mean Ratio (and 90%CI) | At steady state, on the sixth planned treatment day
  AUCτ,ss Geometric Mean Ratio for gemigliptin when administered concomitanty with metformin (test) to its administration alone (reference)

SECONDARY OUTCOMES:
Gemigliptin Cmax,ss Geometric Mean Ratio (and 90%CI) | At steady state, on the sixth planned treatment day
  Cmax,ss Geometric Mean Ratio for gemigliptin when administered concomitanty with metformin (test) to its administration alone (reference)
Metformin AUCτ,ss Geometric Mean Ratio (and 90%CI) | At steady state, on the sixth planned treatment day
  AUCτ,ss Geometric Mean Ratio for metformin when administered concomitanty with metformin (test) to its administration alone (reference)
Metformin Cmax,ss Geometric Mean Ratio (and 90%CI) | At steady state, on the sixth planned treatment day
  Cmax,ss Geometric Mean Ratio for metformin when administered concomitanty with metformin (test) to its administration alone (reference)
Ctrough,ss | At steady state, on the sixth planned treatment day
  Lowest plasma concentration prior to the next dose administration at steady state
Aeτ,ss | At steady state, on the sixth planned treatment day
  cumulative amount of drug excreted in the urine during a dosing interval
CLss/F | At steady state, on the sixth planned treatment day
  Apparent drug clearance
CLR,ss | At steady state, on the sixth planned treatment day
  Renal drug clearance
MR | At steady state, on the sixth planned treatment day
  Metabolic ratio
Tmax | At steady state, on the sixth planned treatment day
  Time to maximum plasma concentration at steady state

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events | From the first pre-treatment admission date, trough the 39 days required for completion of the planned treatment/sampling and washout periods up to and including the post-study safety visit, conducted at study day 44
  Incidence of adverse events occuring during the exposure to the study medications

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Conde-Carmona, MD, Study Chair — Específicos Stendhal S.A. de C.V.
Locations (1):
- Unidad de Farmacología Clínica de la Facultad de Medicina de la Universidad Nacional Autónoma de México, Nezahualcóyotl, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No
No formal plan has been established since at the time the study was conducted no consent was obtained from the subjects to share their individual data for research purposes different from those specifically defined in the study protocol

REFERENCES:
- [Background] Kim SH, Jung E, Yoon MK, Kwon OH, Hwang DM, Kim DW, Kim J, Lee SM, Yim HJ. Pharmacological profiles of gemigliptin (LC15-0444), a novel dipeptidyl peptidase-4 inhibitor, in vitro and in vivo. Eur J Pharmacol. 2016 Oct 5;788:54-64. doi: 10.1016/j.ejphar.2016.06.016. Epub 2016 Jun 11. PMID 27298192
- [Background] Lim KS, Kim JR, Choi YJ, Shin KH, Kim KP, Hong JH, Cho JY, Shin HS, Yu KS, Shin SG, Kwon OH, Hwang DM, Kim JA, Jang IJ. Pharmacokinetics, pharmacodynamics, and tolerability of the dipeptidyl peptidase IV inhibitor LC15-0444 in healthy Korean men: a dose-block-randomized, double-blind, placebo-controlled, ascending single-dose, Phase I study. Clin Ther. 2008 Oct;30(10):1817-30. doi: 10.1016/j.clinthera.2008.10.013. PMID 19014837
- [Background] Lim KS, Cho JY, Kim BH, Kim JR, Kim HS, Kim DK, Kim SH, Yim HJ, Lee SH, Shin SG, Jang IJ, Yu KS. Pharmacokinetics and pharmacodynamics of LC15-0444, a novel dipeptidyl peptidase IV inhibitor, after multiple dosing in healthy volunteers. Br J Clin Pharmacol. 2009 Dec;68(6):883-90. doi: 10.1111/j.1365-2125.2009.03376.x. PMID 20002082
- [Background] Kim N, Patrick L, Mair S, Stevens L, Ford G, Birks V, Lee SH. Absorption, metabolism and excretion of [14C]gemigliptin, a novel dipeptidyl peptidase 4 inhibitor, in humans. Xenobiotica. 2014 Jun;44(6):522-30. doi: 10.3109/00498254.2013.865856. Epub 2013 Dec 4. PMID 24304170
- [Background] Ingelman-Sundberg M, Sim SC, Gomez A, Rodriguez-Antona C. Influence of cytochrome P450 polymorphisms on drug therapies: pharmacogenetic, pharmacoepigenetic and clinical aspects. Pharmacol Ther. 2007 Dec;116(3):496-526. doi: 10.1016/j.pharmthera.2007.09.004. Epub 2007 Oct 9. PMID 18001838
- [Background] Zanger UM, Schwab M. Cytochrome P450 enzymes in drug metabolism: regulation of gene expression, enzyme activities, and impact of genetic variation. Pharmacol Ther. 2013 Apr;138(1):103-41. doi: 10.1016/j.pharmthera.2012.12.007. Epub 2013 Jan 16. PMID 23333322
- [Background] Reyes-Hernandez OD, Lares-Asseff I, Sosa-Macias M, Vega L, Albores A, Elizondo G. A comparative study of CYP3A4 polymorphisms in Mexican Amerindian and Mestizo populations. Pharmacology. 2008;81(2):97-103. doi: 10.1159/000109983. Epub 2007 Oct 19. PMID 17952011
- [Background] Shin D, Cho YM, Lee S, Lim KS, Kim JA, Ahn JY, Cho JY, Lee H, Jang IJ, Yu KS. Pharmacokinetic and pharmacodynamic interaction between gemigliptin and metformin in healthy subjects. Clin Drug Investig. 2014 Jun;34(6):383-93. doi: 10.1007/s40261-014-0184-3. PMID 24627290
- [Derived] Conde-Carmona I, Garcia-Medina S, Jimenez-Vargas JM, Martinez-Munoz A, Lee SH. Pharmacokinetic Interactions Between Gemigliptin and Metformin, and Potential Differences in the Pharmacokinetic Profile of Gemigliptin Between the Mexican and Korean Populations: A Randomized, Open-label Study in Healthy Mexican Volunteers. Clin Ther. 2018 Oct;40(10):1729-1740. doi: 10.1016/j.clinthera.2018.08.015. Epub 2018 Sep 22. PMID 30249366